CLINICAL TRIAL: NCT07141888
Title: The Effects of a Novel Probiotic Food Supplement in Hyperuricaemia - Towards Development of an Individualised Treatment Strategy
Brief Title: The Effects of a Probiotic Food Supplement in Hyperuricaemia
Acronym: Bugs4U-PoC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Julia König, PhD, Associate professor, PhD, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-04358-01
Record Dates: First submitted 2025-08-15; First posted 2025-08-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hyperuricemia With or Without Gout
MeSH Terms: interventions — Probiotics; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo - no active ingredients (Placebo Comparator): No active ingredients
  Interventions: Dietary Supplement: Placebo (no active ingredient)
- Probiotic product (Experimental): Product contains two probiotic strains
  Interventions: Dietary Supplement: Probiotics
- Probiotic product plus fibre (Experimental): Product contains two probiotic strains and a fibre (beta-glucan)
  Interventions: Dietary Supplement: Probiotics plus fibre

INTERVENTIONS:
Dietary Supplement: Placebo (no active ingredient) — Placebo product containing the same ingredients as the active intervention but without the active compounds
  Arms: Placebo - no active ingredients
Dietary Supplement: Probiotics — Product contains two probiotic strains
  Arms: Probiotic product
Dietary Supplement: Probiotics plus fibre — Product contains two probiotic strains plus a fibre (beta-glucan)
  Arms: Probiotic product plus fibre

SUMMARY:
The overall aim of the project is to determine whether a daily intake of health-promoting bacteria, known as probiotics, with or without a dietary fiber, affects uric acid levels in individuals with elevated levels of uric acid in the blood (hyperuricemia). Additionally, the project will investigate which individuals benefit from this dietary supplement and which do not, based on factors such as gut microbiota composition and function, dietary habits, genetic factors, and inflammatory status. The ultimate goal is to develop a personalized therapy for hyperuricemia.

At the beginning of the study, blood samples will be taken to determine uric acid levels and 99 individuals with hyperuricemia will be invited to participate in a 6-week intervention study with daily intake of dietary supplements. To examine the effect of the supplement on various health variables, blood, urine, stool, and breath samples will be collected on several occasions.

To better understand the underlying factors of hyperuricemia, questionnaire data and results from biological will be compared between participants with normal versus elevated uric acid levels. Furthermore, different outcome parameters from questionnaires and samples before and after supplement intake will be compared. In addition, various methods for estimating dietary intake will be investigated and compared with each other.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-related procedures
2. Age 18-80 years old
3. BMI range 17.5-40 kg/m2
4. Blood uric acid above 405 μmol/l (6.8 mg/dl)
5. Willing to abstain from regular consumption of probiotic supplements or food products containing probiotic bacteria (including fermented food and beverages) during the study
6. Willing to abstain from regular consumption of supplements and medications known to alter gastrointestinal function or inflammatory status during the study

Exclusion Criteria:

1. Recent (within last month) episode of gout
2. Diagnosis of type 1 diabetes
3. Diagnosed inflammatory bowel disease (IBD)
4. Current diagnosis of psychiatric disease/s or syndromes
5. Current diagnosis of neurodegenerative disease
6. Current pregnancy or breastfeeding
7. History of complicated gastrointestinal surgery
8. (Partial) resection of the small intestine or colon
9. Regular use of urate-lowering treatment (apart from allopurinol) in the month prior to inclusion
10. Oral or intravenous administration of antibiotics and/or corticosteroids in the 4 months prior to inclusion
11. Regular use of any non-steroidal anti-inflammatory drug (NSAID) during the last month prior to inclusion (apart from low-dose acetylsalicylic acid)
12. Consumption of more than 9 standard glasses of alcohol-containing drinks per week and/or more than 4 standard glasses per occasion
13. Regular use of probiotic or prebiotic supplementation in the month prior to inclusion
14. Any condition or intake of medication which could substantially interfere with the outcome of the study, as decided by the principal investigator's discretion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Effect of a 6-week intake of a probiotic product on blood urate levels in hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood urate levels in the probiotic intervention arm after six weeks will be compared to the levels in the placebo arm

SECONDARY OUTCOMES:
Effect of a 3-week intake of a probiotic product on blood urate levels in hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected blood urate levels in the probiotic intervention arm after three weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on blood urate levels in hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected blood urate levels in the probiotic plus fibre intervention arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on blood urate levels in hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood urate levels in the probiotic plus fibre intervention arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on blood urate-related metabolites in hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected blood urate-related metabolite levels in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on blood urate-related metabolites in hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood urate-related metabolite levels in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on blood urate-related metabolites in hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected blood urate-related metabolite levels in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on blood urate-related metabolites in hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood urate-related metabolite levels in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on blood urate-related enzymes in hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected blood urate-related enzyme levels in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on blood urate-related enzymes in hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood urate-related enzyme levels in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on blood urate-related enzymes in hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood urate-related enzyme levels in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on blood urate-related enzymes in hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood urate-related enzyme levels in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on urate-related metabolites in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related metabolite levels in stool samples in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on urate-related metabolites in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related metabolite levels in stool samples in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on urate-related metabolites in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related metabolite levels in stool samples in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on urate-related metabolites in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related metabolite levels in stool samples in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on urate-related enzymes in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related enzyme levels in stool samples in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on urate-related enzymes in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related enzymes levels in stool samples in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on urate-related enzymes in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related enzyme levels in stool samples in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on urate-related enzymes in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related enzyme levels in stool samples in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on urate-related enzymes in urine of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related enzymes levels in urine samples in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on urate-related enzymes in urine of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related enzymes levels in urine samples in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on urate-related enzymes in urine of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related enzymes levels in urine samples in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on urate-related enzymes in urine of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related enzymes levels in urine samples in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on inflammation markers in blood of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected inflammation markers in blood samples in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on inflammation markers in blood of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected inflammation markers in blood samples in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on inflammation markers in blood of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected inflammation markers in blood samples in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on inflammation markers in blood of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected inflammation markers in blood samples in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on inflammation markers in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected inflammation markers in stool samples in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on inflammation markers in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected inflammation markers in stool samples in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on inflammation markers in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected inflammation markers in stool samples in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on inflammation markers in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected inflammation markers in stool samples in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on blood creatinine levels of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected blood creatinine levels (eGFR - estimated glomerular filtration rate) in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on blood creatinine levels of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood creatinine levels (eGFR - estimated glomerular filtration rate) in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on blood creatinine levels of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected blood creatinine levels (eGFR - estimated glomerular filtration rate) in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on blood creatinine levels of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected blood creatinine levels (eGFR - estimated glomerular filtration rate) in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on urine creatinine levels of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urine creatinine levels in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on urine creatinine levels of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urine creatinine levels in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on urine creatinine levels of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urine creatinine levels in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on urine creatinine levels of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urine creatinine levels in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on urate levels in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate levels in stool samples of the probiotic intervention arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on urate levels in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate levels in stool samples of the probiotic intervention arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on urate levels in stool of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate levels in stool samples of the probiotic plus fibre intervention arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on urate levels in stool of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate levels in stool samples of the probiotic plus fibre intervention arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on urate levels in urine of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate levels in urine samples of the probiotic intervention arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on urate levels in urine of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate levels in urine samples of the probiotic intervention arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on urate levels in urine of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate levels in urine samples of the probiotic plus fibre intervention arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on urate levels in urine of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate levels in urine samples of the probiotic plus fibre intervention arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product on urate-related metabolites in urine of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related metabolite levels in urine samples in the probiotic arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product on urate-related metabolites in urine of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related metabolite levels in urine samples in the probiotic arm after six weeks will be compared to the levels in the placebo arm
Effect of a 3-week intake of a probiotic product in combination with a fibre on urate-related metabolites in urine of hyperuricaemic individuals compared to placebo | 3 weeks
  Baseline-corrected urate-related metabolite levels in urine samples in the probiotic plus fibre arm after three weeks will be compared to the levels in the placebo arm
Effect of a 6-week intake of a probiotic product in combination with a fibre on urate-related metabolites in urine of hyperuricaemic individuals compared to placebo | 6 weeks
  Baseline-corrected urate-related metabolite levels in urine samples in the probiotic plus fibre arm after six weeks will be compared to the levels in the placebo arm

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
According to Swedish ethics regulations, IPD cannot be shared without an approved ethics application from the National Swedish Ethics Authority. An ethical permit can only be obtained for research being conducted within Sweden.